CLINICAL TRIAL: NCT04305314
Title: Surgical Treatment of Colorectal Cancer: Analysis of the Influence of an Enhanced Recovery Protocol on Long-term Oncological Outcomes.
Brief Title: Long-term Enlarged Survival After an Enhanced Recovery Protocol (LESAS).
Acronym: LESAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Sponsor
Other Study IDs: GERMFIS2020
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Major Surgery
MeSH Terms: interventions — placental ribonuclease inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: PRI > 70%: Compliance with the Enhanced Revovery protocol higher than 70%
  Interventions: Other: PRI (Enhanced Recovery after surgery protocol)
- Group 2: PRI < 70%: Compliance with the Enhanced Revovery protocol lower than 70%

INTERVENTIONS:
Other: PRI (Enhanced Recovery after surgery protocol) — Standard use of Spanish perioperative guidelines (PRI)
  Groups: Group 1: PRI > 70%

SUMMARY:
The main objective of this study is to analyze the impact on three years survival of an enhanced recovery program (PRI) after radical surgery for colorectal cancer. As secondary objectives, we propose to analyze the weight of each of the predefined items in the oncological results as well as the quality of life.

We design a multicentric prospective cohort study in people older than 18 years who are going to be operated on for colorectal cancer. 12 hospitals are being selected due to have a PRI implanted according to the RICA pathway published by the Spanish National Health Service. As stated by the literature, the intervention group will be formed for those hospitals with a minimum implementation level of 70% of the PRI and the control group will be the centers that do not reach this level of implementation. Compliance will be studied with 21 key performance indicators and results are analyzed with cancer survival indicators: Overall survival, cancer-specific survival and relapse-free survival). We will also study the time to recurrence, perioperative morbi-mortality, hospital stay and quality of life with the EQ-5D validated questionary.

To create comparable treatment and control groups, the Propensity Index method will be used. To study each variable, multivariate regression will be used. Kaplan-Meier will be used for survival and the log-rank test for comparisons. Significance will be considered if p <0.05 (two tails).

DETAILED DESCRIPTION:
Subjects of study (inclusion criteria): All patients over 18 years of age who will be operated on a scheduled basis for colorectal cancer within an intensified recovery program (PRI) and who do not present any exclusion criteria.

Exclusion Criteria: - Urgent surgery; -Existence of other concomitant surgical processes; -Patients diagnosed in stage IV cancer; -Patients who refuse to participate.

Participating hospitals: Selected for their interest in intensified recovery and for having established a multidisciplinary team with the program (PRI) for colorectal surgery recommended by the Spanish Ministry of Health. Each center will select from the multidisciplinary team the researchers who will be part of this project as collaborators, ideally the facilitators of the PRI program in that center.

Variables: Patients will be recruited by local researchers from the Anesthesiology and Resuscitation and/or General Surgery services of each participating center before performing the surgical intervention. Informed consent will be requested from all subjects who voluntarily participate in the study.

1. Compliance: As we have commented before and according to the literature, we will define a hospital with an intensified recovery program (PRI) that has a consensus protocol, based on evidence, multidisciplinary, with the support of the center (management) and that has fulfilled more than 70% of the protocol (annex 1) according to the process indicators. The rest of the hospitals will be considered a non-PRI hospital.
2. Demography: Age, sex, BMI, smoking and fitness level of the American Society of Anesthesiologists (ASA). BMI in the surgical indication. Blood transfusion.
3. Comorbidities: Presence of hypertension, diabetes mellitus, coronary artery disease, heart failure, cirrhosis, stroke or transient ischemic attack, COPD / Asthma, atrial fibrillation, heart failure, OSAS. Anemia
4. Related to Surgery and Treatment: Date IQ. Surgical procedure, approach, duration of surgery, estimated bleeding. Curative surgery (R0) or non-R0 (R1-R2). Adjuvant chemotherapy Adjuvant radiotherapy Perioperative transfusion.
5. Variables related to staging: Tumor typology. Growth pattern. Degree of differentiation. Presence of Vascular / lymphatic / perineural invasion / Satellites. Margin affectation. Seal ring cells. K-ras. T tumor piece. No tumor piece. Tumor m. Tumor stage according to AJCC classification.
6. Related to the follow-up:

In-hospital complications at 60 days of follow-up that will be recorded are: surgical complications, infectious complications, cardiovascular complications and other types of complications. Each complication will be classified as mild, moderate or severe. The Clavien-Dindo classification will also be used. Perioperative mortality: The number and percentage of deaths within 60 days of surgery. Hospital Stay: hospital stay is defined as the duration in days from the date of admission to hospital discharge. Quality of life according to the EuroQol Five questionnaire. (EQ-5D).

Overall mortality: The number and percentage of deaths occurred since the intervention until the end of the follow-up period. Overall survival: patients alive from surgery to the last control. Disease-free survival: number of patients alive and without cancer recurrence from the intervention period until the end of follow-up.

Disease recurrence: detected by CT or FCC, from the day of the intervention until the end of the follow-up.

Patient Follow-up Plan: 5 years after surgery. Data collection: The data will be collected in individual hospitals on a paper CRD for each patient recruited. This will include patient identification data in order to allow monitoring of clinical results. The data will be encoded by generating a unique numerical code and transcribed by local researchers in a database using an electronic CRD (eCRD). The data collection platform used will be Castor EDC https://www.castoredc.com/. Castor EDC complies with all applicable laws and regulations: good clinical practice (GCP), 21 CFR Part 11, EU Annex 11 and the European Data Protection Directive. Each patient will only be identified in the electronic CRD by their numerical code. In each center a list of patients will be used to match the identification codes of the individual patients' database in order to record the clinical results and provide any of the missing data. All identifiable data collected, processed and stored for the purposes of the project will be kept confidential at all times and will comply with the guidelines of Good Clinical Practice for Research (GCP) and the General Data Protection Regulation (GDPR) (Regulation (EU) ) 2016/679).

Data analysis: Sample size: understanding, according to the literature, that only 60% of the centers with a PRI achieve more than 70% of compliance, we consider the scenario of 6 PRI and 4 non-PRI centers adequate among the 10 who collaborate in this research project. Estimating a difference in overall survival between centers around 10% (65% vs. 75%), with a power of 80%, a 95% confidence and 5% of possible losses, a minimum sample size of 366 is estimated patients in each group (732 patients in total). For the study of survival, only patients with a minimum follow-up of two years (first 12 months of the study) will be considered. However, they will continue to be recruited until the end of the three years for the study of secondary objectives.

Understanding that the main objective, study of survival, may be subject to inherent aspects of each center, independent of the intervention, it is necessary to create comparable treatment and control groups for which the Propensity Score (Propensity Score Matching) method will be used. A descriptive analysis of the data will be carried out: Qualitative variables will be presented by frequency distribution of the percentages of each category. The quantitative variables studied will be explored with the Kolmogorov - Smirnov conformity test. Bivariate Analysis Comparison between variables (factors): The association between the factors will be investigated by hypothesis contrast tests, with comparison of proportions when both variables are qualitative (chi square, Fisher's exact test), mean comparisons when one of them is quantitative (Student's t, ANOVA, and if they do not follow the normal distribution, the Mann-Whitney U test or the Kruskall-Wallis test) and bivariate correlations (Coef. Pearson Correlation) when both are quantitative or, if the conditions are not met of application, the Spearman correlation. For comparisons in related samples when one of them is quantitative, Student's t-test and/or ANOVA will be used for repeated measurements and Wilcoxon or Friedman's test when do not follow normal distribution). Multivariate analysis: To study the relationship of each variable controlling the possible effect caused by third variables. The analysis will be completed using multivariate regression models. Survival analyzes will be performed using the Kaplan-Meier method for survival comparisons the log-rank test will be used. The effects will be considered significant if p <0.05.

Monitoring and audit: The data collection documents will be audited to ensure that study activities are carried out in accordance with the protocol, good clinical practice and applicable regulatory requirements. In the participating hospitals, local study documents can be selected for local auditing. The quality of the data will be audited.

Limitations of the study: Those of a prospective non-randomized study. Difficulty in recruiting patients for potential structural or multidisciplinary team problems. Inappropriate number of patients in any of the arms due to a very high or very low level of compliance.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age who will be operated on a scheduled basis for colorectal cancer

Exclusion Criteria:

* - Urgent surgery; -Existence of other concomitant surgical processes; -Patients diagnosed in stage IV cancer; -Patients who refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter prospective observational cohort study in patients who meet inclusion criteria (18 years of age who will be operated on a scheduled basis for colorectal cancer ) in participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  patients alive from surgery to the last control
Disease-free survival | 5 years
  number of patients alive and without cancer recurrence from the intervention period until the end of follow-up
Disease recurrence | 5 years
  detected from the day of the intervention until the end of follow-up

SECONDARY OUTCOMES:
Compliance of individual items of the protocol | 5 years
  To evaluate the relationship between adherence to the protocol and 5-year survival
Quality of Life (QOL) | 5 years
  Quality of life according to the EuroQol (EQ-5D)
Patient reported outcoms (PROs) | 5 years
  According to EuroQol (EQ-5D) and self-completed disease-specific PROM questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Ramirez, Prof., Principal Investigator — Universidad de Zaragoza
Locations (12):
- Spain (12):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital de la Ribera, Alzira
  - Hospital de Barbastro, Barbastro
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Jiménez Diaz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Complejo Asistencial Universitario de Palencia, Palencia
  - Hospital General de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramirez-Rodriguez JM, Martinez-Ubieto J, Munoz-Rodes JL, Rodriguez-Fraile JR, Garcia-Erce JA, Blanco-Gonzalez J, Del Valle-Hernandez E, Abad-Gurumeta A, Centeno-Robles E, Martinez-Perez C, Leon-Arellano M, Echazarreta-Gallego E, Elia-Guedea M, Pascual-Bellosta A, Miranda-Tauler E, Manuel-Vazquez A, Balen-Rivera E, Alvarez-Martinez D, Perez-Pena J, Abad-Motos A, Redondo-Villahoz E, Biosta-Perez E, Guadalajara-Labajo H, Ripolles-Melchor J, Latre-Saso C, Cordoba-Diaz de Laspra E, Sanchez-Guillen L, Cabellos-Olivares M, Longas-Valien J, Ortega-Lucea S, Ocon-Breton J, Arroyo-Sebastian A, Garcia-Olmo D. Surgical treatment for colorectal cancer: analysis of the influence of an enhanced recovery programme on long-term oncological outcomes-a study protocol for a prospective, multicentre, observational cohort study. BMJ Open. 2020 Oct 27;10(10):e040316. doi: 10.1136/bmjopen-2020-040316. PMID 33109675